CLINICAL TRIAL: NCT06251141
Title: Effectiveness of Gum Health Gel in Minimizing Post Operative Sequelae Associated With the Surgical Removal of Impacted Mandibular Third Molars
Brief Title: Gum Health Gel in Post Extraction Sockets
Acronym: Gum Health gel
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Baghdad (Other)
Responsible Party: Principal Investigator, Dhuha Ali Bardan, Principal investigator, University of Baghdad
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 894124
Record Dates: First submitted 2024-01-23; First posted 2024-02-09 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2024-02

CONDITIONS: Impacted Third Molar Tooth
MeSH Terms: interventions — Vaginal Creams, Foams, and Jellies

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group gum Health gel (Active Comparator): Study group we fill the sockets with gel foam immersed with Gum Health gel
  Interventions: Procedure: Gum Health gel
- Control group gel foam (Placebo Comparator): Control group we fill the sockets with gel foam only
  Interventions: Procedure: Gel foam

INTERVENTIONS:
Procedure: Gum Health gel — Extraction of impacted mandibular third molars under local anaesthesia and irrigating the socket with normal saline, and filling the socket with the Gum Health gel
  Arms: Study group gum Health gel
Procedure: Gel foam — Extraction of impacted mandibular third molars under local anaesthesia and irrigating the socket
  Arms: Control group gel foam

SUMMARY:
This research studies the effectiveness of the Gum Health gel in minimizing post operative sequelae associated with the surgical removal of impacted mandibular third molars

DETAILED DESCRIPTION:
This research studies the effectiveness of the Gum Health gel in minimizing post operative sequelae associated with the surgical removal of impacted mandibular third molars which includes pain , swelling and trismus

ELIGIBILITY:
Inclusion Criteria: Horizontal and mesioangular impaction in healthy patients older than 18 years old -

Exclusion Criteria:any medically compromised patient and the presence of any infection

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2024-02-15 (Actual); Primary Completion 2024-08-19 (Estimated); Study Completion 2024-09-19 (Estimated)

PRIMARY OUTCOMES:
Decrease of Pain | One week
  Pain with Visual analog scale
Increase Soft tissue healing | One week
  Soft tissue healing with Early wound healing scale
Decrease in Trismus | One week
  Trismus with Maximum-interincisal- opening (MIO) thatimillimeters
Decrease of Swelling | One week
  Swelling withGrades of swelling

CONTACTS AND LOCATIONS:
Locations (1):
- Collage of dentistry/ university of baghdad, Baghdad, Iraq